CLINICAL TRIAL: NCT06113588
Title: Improving Transition of Care in Type 1 Diabetes Mellitus: A Collaborative Approach
Brief Title: Transition of Care in Type 1 Diabetes Mellitus
Status: Enrolling by invitation | Type: Observational
Sponsor: Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Principal Investigator, Shihab Hameed, Principal Investigator, Northern Sydney and Central Coast Area Health Service
Other Study IDs: 2022/ETH02412
Record Dates: First submitted 2023-06-21; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Transition; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: Patients with type 1 diabetes mellitus known to Royal North Shore Hospital, who underwent transition from paediatric to adult health care from 1st January 2020-8th June 2023
- Prospective cohort: Patients with type 1 diabetes mellitus known to Royal North Shore Hospital, undergoing transition from paediatric to adult health care, from 9th June 2023 onwards

SUMMARY:
This research project seeks to address the question of how to improve the transition of patients with type 1 diabetes mellitus from the paediatric to the adult health service at RNSH and Mona Vale Community Health Centre (seeking the perspectives of patients, families, and staff)?

DETAILED DESCRIPTION:
There are significant limitations in the literature relating to transition from paediatric to adult healthcare.

In healthcare, transition describes the purposeful process of planning and moving from paediatric to adult services and usually occurs in adolescence (in itself a time of rapid physical, cognitive and psychosocial growth between childhood and adulthood). The available evidence within the literature to guide this process of transition is often limited and additional evidence to guide clinical practice is required. Although reports within the literature vary, it is known that up to 50% of young adults with an endocrine disorder are lost to follow-up after transition to adult health services. Even if the young person attends the adult service, they may have poor health outcomes related to inability to self-manage their condition, particularly if it is a chronic disease requiring significant daily intervention by the patient, such as in type 1 diabetes mellitus.

Type 1 diabetes mellitus is a life-long condition characterised by autoimmune-mediated destruction of pancreatic β-cells, almost always resulting in absolute insulin deficiency. As a result, patients are required to perform lifelong intensive glucose monitoring and insulin administration. These intensive insulin regimens require an enormous amount of attention and effort on the part of the young person with diabetes and their family, but dramatically reduce their rates of micro- and macro-vascular complications, such as blindness, kidney failure, heart attack and stroke. Evidence for this 'legacy effect' - the long-term clinical benefits of early intensive insulin treatment - are provided through studies including the EDIC (Epidemiology of Diabetes Interventions and Complications) study which undertook long-term follow up of the Diabetes Control and Complications Trial (DCCT). The DCCT, conducted from 1983-1989, randomised 1441 participants with new or recently-diagnosed type 1 diabetes to receive either intensive insulin therapy or standard therapy. The DCCT/EDIC study ultimately recommended maintaining patients' glucose levels as close to the normal range as safely possible, with intensive insulin therapy and monitoring.

Glycaemic control and transition in adolescents with type 1 diabetes mellitus has its own specific challenges. Across all age groups, adolescents are currently the farthest from achieving good glycaemic control (a HbA1c goal of <58 mmol/mol or 7.0%). The factors contributing to this may include hormonal changes during puberty, psycho-social challenges and decreased adherence to insulin therapy regimens.

Appropriate transition of patients with type 1 diabetes from paediatric to adult health care thus needs to take a holistic approach to the individual patient which addresses these factors and which is centred on individual patients' developmental stages and circumstances.

The local transition process at Royal North Shore Hospital has future potential At Royal North Shore Hospital, there is a structured transition process underpinned by the transition policy. However, initial analysis indicates that patients are missing appointments and education, and being lost to follow-up. There is accordingly a pressing need for analysis of the transition process and its outcomes.

Within the current literature, evaluation measures to assess patients' diabetes self-management and transition readiness (including glucose monitoring, insulin and food regulation, exercise, and emergency preparedness) frequently rely on patient self-report and emphasise knowledge and practical skills in diabetes care.

This research will provide additional insights from the patient's family and from treating staff as well as explore self-efficacy (the individual's belief in their capacity to execute behaviours) which are often poorly studied in transition research. It is anticipated that this will provide a comprehensive picture of areas in which patients' efficacy, transition readiness, knowledge and diabetes-related distress can have tailored support provided in an individualised way.

This research project will utilise the following questionnaires, with access for all participants via a QR code using Northern Sydney Local Health District (NSLHD) REDCap (a secure, web-based application for building and managing online surveys and databases).

1. A modified READDY tool assessing transition readiness and self-efficacy - with versions that can be answered separately by the patient, the patient's family member, and the patient's healthcare professional.
2. Diabetes knowledge questionnaire - with versions that can be answered separately by the patient and patient's family member
3. Diabetes distress questionnaire - with versions that can be answered separately by the patient and the patient's family member
4. Evaluation of the transition process - with versions that can be answered separately by patient, patient's family member and staff member

ELIGIBILITY:
Inclusion Criteria:

Adolescents who have an existing diagnosis of type 1 diabetes mellitus and who underwent (in 2020 to 8th June, 2023) or who are undergoing (from 9th June, 2023 and subsequent cohorts) transition from paediatric care to adult health care at Royal North Shore Hospital and Mona Vale Community Health Centre. Adolescents with type 1 diabetes will be 16 years or older

A family member or caregiver of the participant of the adolescent patient with type 1 diabetes mellitus

A staff member who is a member of the patient's treating diabetes team within the paediatric diabetes service (first study visit and second study visit) and young adult diabetes service (third study visit)

Exclusion Criteria:

There are no specific exclusion criteria

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 1 diabetes mellitus meeting inclusion criteria, above
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-06-09 (Estimated); Study Completion 2028-06-09 (Estimated)

PRIMARY OUTCOMES:
Patient self-efficacy (patient, family and staff member) relating to diabetes | From 9th June, 2023, ongoing for initial period of 5 years with interim sequential reviews
  From prospective questionnaires, with higher scores indicative of higher self-efficacy
Diabetes knowledge questionnaire (patient and family member) | From 9th June, 2023, ongoing for initial period of 5 years with interim sequential reviews
  From prospective questionnaires, with a single correct answer per question
Diabetes-related distress (patient and family member) | From 9th June, 2023, ongoing for initial period of 5 years with interim sequential reviews
  From prospective questionnaires, with higher scores indicative of higher distress levels

SECONDARY OUTCOMES:
Patient medical outcomes | From 9th June, 2023, ongoing for initial period of up to 5 years with interim sequential reviews
  HbA1c (%) over time
Patient medical outcomes | From 9th June, 2023, ongoing for initial period of up to 5 years with interim sequential reviews
  Frequency (number) of emergency department presentations
Patient medical outcomes | From 9th June, 2023, ongoing for initial period of up to 5 years with interim sequential reviews
  Percentage of patients developing diabetes complications

CONTACTS AND LOCATIONS:
Overall Officials: Shihab Hameed, MBBS, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Royal North Shore Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No